CLINICAL TRIAL: NCT04409548
Title: Preoperative and Postoperative Spatiotemporal Gait Parameters and Gait Asymmetry in Patients With Lumbar Disc Herniation: a Prospective, Cross-sectional Study
Brief Title: The Spatiotemporal Gait Parameters in LDH Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Collaborators: Bahçeşehir University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bahçeşehir University
Record Dates: First submitted 2020-05-12; First posted 2020-06-01 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2020-05

CONDITIONS: Lumbar Disc Herniation; Pain
Keywords: Pain; Gait analysis; Lumbar Disc Herniation; Spatiotemporal gait parameters; Gait asymmetry
MeSH Terms: conditions — Intervertebral Disc Displacement; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lumbar Disc Hernaition Group (Active Comparator): The number of participants in this group is anticipated to be 153. The pain intensity of the patients was recorded by a Visual Analog Scale (VAS) immediately before performing the analysis. The patients were asked to continuously walk barefoot for ten times as straight as possible without any assistance on the Win-Track platform within the same day.
  Interventions: Other: All of the spatial and Temporal Gait parameters
- Healthy Control Group (Active Comparator): The number of participants in this group is anticipated to be 54. The participants were asked to continuously walk barefoot for ten times as straight as possible without any assistance on the Win-Track platform within the same day.
  Interventions: Other: All of the spatial and Temporal Gait parameters
- Preoperative and Postoperative Group (Active Comparator): The number of participants in this group is anticipated to be 59. The patients were asked to continuously walk barefoot for ten times as straight as possible without any assistance on the Win-Track platform within the same day, before and 15 days after surgery.
  Interventions: Other: All of the spatial and Temporal Gait parameters

INTERVENTIONS:
Other: All of the spatial and Temporal Gait parameters

SUMMARY:
The aim of this study was to assessment on the interaction of spatial and temporal gait parameters and gait asymmetry in patients with Lumbar Disc Herniation (LDH) before and 15 days after surgery.

DETAILED DESCRIPTION:
The participants were divided into LDH and healthy control groups. The analysis of the spatiotemporal gait parameters was performed using the "Win-Track" gait analysis platform system for two groups. In addition, the analysis of spatiotemporal gait parameters of 60 participants who had the planned lumbar discectomy surgery, was tested before and 15 days after surgery. The pain intensity of the patients was recorded by the Visual Analog Scale (VAS) immediately before performing the analysis. After then participants completed ten passes on the "Win-Track" Gait Analysis Platform at their self-selected walking speed. The arithmetic mean of the three flawless walking data was used for analysis. The gait symmetry index was used to calculate the walking asymmetry.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who were diagnosed with LDH by a specialist;
* Patients had a medical history and proven by MRI with more or less evidence of degenerative lumbar disc;
* Aged between 25-80 years old;
* Pain symptom on the lumbal area or lower extremity.

Exclusion Criteria:

* Patients who have previously received surgery or physical therapy treatment;
* Having congenital deformity in the spine or lower extremity;
* History of spinal surgery or other diseases affecting gait;
* Pregnancy;
* Situations that may cause gait balance problems;
* Using assistive gait appliance.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | The pain intensity of the patients was recorded immediately before performing the analysis.
  Pain intensity was obtained using a Visual Analog Scale (VAS). VAS is usually a horizontal line, 10 cm in length, anchored by word descriptors at each end with "No Pain" (score of zero) on the left side up to "pain as bad as it could be" or the "worst imaginable pain" (Score of 100 [100-mm scale]) on the right side. The patient was asked to mark the line point that represented his or her current pain.
Step length (cm) | Changes from the step length at 2 weeks
  Step length is the distance between the heel contact point of one foot and that of the other foot. The step length (cm) was recorded separately for both extremities.
Gait cycle length (cm) | Changes from the gait cycle length at 2 weeks
  Gait cycle length is the distance between successive foot contacts of the same limbs. The gait cycle length (cm) was recorded separately for both extremities.
Cadence (step/min) | Changes from the cadence at 2 weeks
  Cadence is the number of steps per minute.
Velocity (cm/s) | Changes from the velocity at 2 weeks
  Velocity is the distance covered in a given period.
Gait cycle duration (seconds) | Changes from the gait cycle duration at 2 weeks
  Gait cycle duration is the time between successive foot contacts of the same limbs. The gait cycle duration (seconds) was recorded separately for both extremities.
Step duration (seconds) | Changes from the step duration at 2 weeks
  Step duration is the time between two consecutive heel strikes. The step duration (seconds) was recorded separately for both extremities.
Double stance duration (seconds) | Changes from the double stance duration at 2 weeks
  Double stance duration is the time over which the body is supported by both legs. The double stance duration (seconds) was recorded separately for both extremities.
Swing duration (seconds) | Changes from the swing duration at 2 weeks
  Swing duration is the time taken for the leg to swing through while the body is in single support on the other leg. The swing duration (seconds) was recorded separately for both extremities.
Gait symmetry | Changes from the gait asymmetry at 2 weeks (preoperative and postoperative).
  Gait symmetry is a coordinated and consistent activity of locomotion between left and right limb during walking.

CONTACTS AND LOCATIONS:
Overall Officials: TUGBA KURU COLAK, Assoc. Prof., Study Director — Marmara University

REFERENCES:
- [Background] Toosizadeh N, Yen TC, Howe C, Dohm M, Mohler J, Najafi B. Gait behaviors as an objective surgical outcome in low back disorders: A systematic review. Clin Biomech (Bristol). 2015 Jul;30(6):528-36. doi: 10.1016/j.clinbiomech.2015.04.005. Epub 2015 Apr 17. PMID 25921552
- [Background] Loske S, Nuesch C, Byrnes KS, Fiebig O, Scharen S, Mundermann A, Netzer C. Decompression surgery improves gait quality in patients with symptomatic lumbar spinal stenosis. Spine J. 2018 Dec;18(12):2195-2204. doi: 10.1016/j.spinee.2018.04.016. Epub 2018 Apr 27. PMID 29709554
- See also: Gait behaviors as an objective surgical outcome in low back disorders: A systematic review. — https://www.ncbi.nlm.nih.gov/pubmed/25921552
- See also: Decompression surgery improves gait quality in patients with symptomatic lumbar spinal stenosis. — https://www.ncbi.nlm.nih.gov/pubmed/?term=Decompression+surgery+improves+gait+quality+in+patients+with+symptomatic+lumbar+spinal+stenosis.

DOCUMENTS (2):
  • Study Protocol (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT04409548/Prot_002.pdf
  • Statistical Analysis Plan (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT04409548/SAP_003.pdf